CLINICAL TRIAL: NCT00442819
Title: Uremic Pruritus, Cytokines and Polymethylmethacrylate Artificial Kidney
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMR95-IRB-79
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Uremia; Pruritus
Keywords: Uremic Pruritus; Cytokines; Polymethylmethacrylate Artificial Kidney; Hemodialysis
MeSH Terms: conditions — Uremia; Pruritus | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Hemodialysis with Polymethylmethacrylate Artificial Kidney

SUMMARY:
Background: Uremic pruritus is one of the common complications in long-term dialysis patients. In general, many factors including xerosis, elevated serum calcium, phosphate, calcium-phosphate product, hyperparathyroidism and inadequate dialysis may contribute to it. Recently, researchers reported that immuno-hypothesis with high serum level of cytokines could be the cause of uremic pruritus. Polymethylmethacrylate (PMMA) artificial kidney (AK) has been reported to adsorb more serum cytokines than other high flux artificial kidneys.

Methods: In July 2006, 30 patients with severe uremic pruritus from 300 chronic hemodialysis patients in a single center entered this prospective study. Their dialyzers were changed to PMMA AK for 4 weeks. The severity of pruritus was evaluated every week using the results of a questionnaire (pruritus score). Laboratory assays including pre-dialysis serum blood urea nitrogen, creatinine, β2-microgblubulin (β2M), calcium, phosphate, intact parathyroid hormone (iPTH), total CO2, ferritin, hematocrit, high sensitivity C-reactive protein (hsCRP), IL-1, IL-2, IL-6, IL-18, TNF-α, KT/V and β2M clearance were measured before and at the end of 4 weeks of PMMA AK use.

Expected Results:To prove the PMMA membrane could improve the uremic pruritus and to reveal the effect of PMMA membrane on serum level of possible factors contributing to uremic pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pruritus (>3 months) were screened using traditional visual analogue scale (VAS) and then scored using a pruritus questionnaire (pruritus scoring system).
* Other inclusion criteria were that patients enrolled should be dialysed for 4 hours, three times a week, with KT/V >1.2, serum albumin> 3.0 mg/dl, hematocrit > 24%, ferritin < 900 ng/ml, phosphate <7 mg/dl, corrected calcium <11 mg/dl, calcium-phosphate product < 70, intact parathyroid hormone (iPTH) <600 pg/ml, and normal serum level of alanine aminotransferase and bilirubin in past 3 months.

Exclusion Criteria:

* Pruritus unrelated to renal failure
* Evidence of malignancy
* Liver cirrhosis diagnosed by echogram or admission within 3 months of the start of the study.

Ages: 26 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-07; Study Completion 2006-09

PRIMARY OUTCOMES:
Improvement of uremic pruritus

SECONDARY OUTCOMES:
Change of serum level of cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Ching Huang, MD, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Result] Kato A, Takita T, Furuhashi M, Takahashi T, Watanabe T, Maruyama Y, Hishida A. Polymethylmethacrylate efficacy in reduction of renal itching in hemodialysis patients: crossover study and role of tumor necrosis factor-alpha. Artif Organs. 2001 Jun;25(6):441-7. doi: 10.1046/j.1525-1594.2001.025006441.x. PMID 11453873